CLINICAL TRIAL: NCT01825785
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 785 in Healthy Men and Postmenopausal Women With Low Bone Mass
Brief Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Romosozumab (AMG 785)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20060221
Record Dates: First submitted 2013-01-25; First posted 2013-04-08 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2019-04

CONDITIONS: Postmenopausal; Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — romosozumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants were randomized to receive matching placebo administered by subcutaneous injection once every 2 weeks (Q2W) or once every 4 weeks (Q4W) for 3 months.
  Interventions: Drug: Placebo
- Romosozumab (Experimental): Participants were randomized to receive romosozumab administered by subcutaneous injection at doses of 1 mg/kg Q2W, 2 mg/kg Q4W, 2 mg/kg Q2W, or 3 mg/kg Q4W for 3 months.
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Administered by subcutaneous injection
  Other Names: AMG 785; EVENITY™
  Arms: Romosozumab
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
The primary objective of this study was to assess the safety, tolerability, and immunogenicity potential of romosozumab following multiple subcutaneous (SC) administrations in healthy men and postmenopausal women with low bone mass.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between 45 to 80 years of age
* Postmenopausal females
* Low bone mineral density, defined by bone mineral density (BMD) T-scores between -1.0 and -2.5, inclusive, for the lumbar spine [L1-L4] or total evaluable vertebrae [if fewer than L1-L4] or total hip)
* 25-hydroxyvitamin D ≥ 20 ng/mL
* Weight ≤ 98 kg (216 lb) and/or height ≤ 196 cm (77 in)

Exclusion Criteria:

* Osteoporosis defined by bone mineral density (BMD) T-scores < -2.5 for the lumbar spine (L1-L4) or total evaluable vertebrae (if fewer than L1-L4) or total hip
* Diagnosed with any condition that would affect bone metabolism
* Previous exposure to AMG 785

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-11-14 (Actual); Primary Completion 2008-12-02 (Actual); Study Completion 2008-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 4 centers in the United States (US) from 14 November 2007 to 2 December 2008.
Pre-assignment Details: Participants were enrolled into 1 of 6 cohorts. In each of cohorts 1 to 4, healthy postmenopausal women were randomized in a 3:1 ratio to receive romosozumab or placebo; In each of cohorts 5 and 6, healthy men were randomized in a 3:1 ratio to receive romosozumab or placebo.
Groups:
- Placebo: Participants were randomized to receive matching placebo administered by subcutaneous injection once every 2 weeks (Q2W) or once every 4 weeks (Q4W).
- Romosozumab 1 mg/kg Q2W in Women; Romosozumab 1 mg/kg Q2W in Men: Participants were randomized to receive 1 mg/kg romosozumab by subcutaneous injection once every 2 weeks for 3 months.
- Romosozumab 2 mg/kg Q4W in Women: Participants were randomized to receive 2 mg/kg romosozumab by subcutaneous injection once every 4 weeks for 3 months.
- Romosozumab 2 mg/kg Q2W in Women: Participants were randomized to receive 2 mg/kg romosozumab by subcutaneous injection once every 2 weeks for 3 months.
- Romosozumab 3 mg/kg Q4W in Women; Romosozumab 3 mg/kg Q4W in Men: Participants were randomized to receive 3 mg/kg romosozumab by subcutaneous injection once every 4 weeks for 3 months.
Period: Overall Study
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 12 | 6 | 6 | 6 | 4 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (5.6) | 56.8 (7.8) | 57.3 (6.6) | 62.5 (8.0) | 54.3 (7.8) | 61.2 (9.0) | 59.3 (12.7) | 58.7 (8.0)
Age, Customized [Count of Participants; unit: Participants]
  18 to 64 years | 11 | 4 | 5 | 4 | 5 | 3 | 4 | 36
  65 to 74 years | 1 | 2 | 1 | 1 | 1 | 3 | 1 | 10
  ≥ 75 years | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 6 | 6 | 6 | 0 | 0 | 32
  Male | 4 | 0 | 0 | 0 | 0 | 6 | 6 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 4 | 5 | 3 | 3 | 3 | 3 | 29
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Hispanic or Latino | 3 | 2 | 1 | 3 | 3 | 3 | 2 | 17
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Serious adverse events were any events that were fatal, were life-threatening (placed the participant at immediate risk of death), required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, were congenital anomalies or birth defects, or were other significant medical hazards.
  Relatedness to investigational product was assessed by the investigator by means of the question: "Is there a reasonable possibility that the event may have been caused by the investigational product?'
Time Frame: 169 days
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Any adverse event | 10 | 6 | 6 | 6 | 5 | 5 | 5
  Serious adverse events | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Treatment-related adverse events | 6 | 1 | 1 | 4 | 3 | 3 | 2
  Treatment-related serious adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Discontinuation due to adverse events | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Death on study | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Developed Antibodies to Romosozumab
Description: All samples were tested for binding anti-romsozumab antibodies using an immunoassay; all antibody-positive samples were further tested in a bioassay to determine if the antibodies were neutralizing.
  Development of antibodies to romosozumab is defined as participants with a negative result at baseline and a positive result at any time postbaseline.
Time Frame: Blood samples for detection of anti-romosozumab antibodies were collected at day 1 (predose) and days 29 (predose), 57 (predose), 85, 113, 141, and 169.
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Binding antibodies | 0 | 2 | 2 | 2 | 3 | 1 | 3
  Neutralizing antibodies | 0 | 1 | 1 | 0 | 0 | 0 | 1

3. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Romosozumab
Description: Serum concentrations of romosozumab were measured by a validated enzyme-linked immunosorbent assay; the lower limit of quantification (LLOQ) was 50 ng/mL.
Time Frame: Q2W dose groups: First dose on days 1 (predose) to 15 (predose); Last dose on days 71 (predose) to 169. Q4W dose groups: First dose on days 1 (predose) to 29 (predose); Last dose on days 57 (predose) to 169.
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be adequately estimated.
Measure: Median (Full Range); unit: days
Arm/Group | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 5 | 6
days
  First dose | 3.0 [2.0 to 5.0] | 3.0 [3.0 to 5.0] | 4.5 [3.0 to 7.0] | 3.0 [3.0 to 5.0] | 3.0 [3.0 to 5.0] | 5.0 [3.0 to 5.0]
  Last dose | 3.0 [3.0 to 5.0] | 3.0 [1.0 to 4.0] | 3.5 [3.0 to 5.0] | 5.0 [2.0 to 7.0] | 3.0 [3.0 to 5.0] | 3.0 [3.0 to 5.0]

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of Romosozumab
Time Frame: as for outcome 3
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be adequately estimated.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 5 | 6
μg/mL
  First dose | 6.80 (1.86) | 15.7 (4.6) | 14.8 (6.0) | 24.5 (6.8) | 8.06 (1.57) | 27.7 (4.2)
  Last dose | 14.2 (4.3) | 16.7 (3.3) | 27.8 (8.4) | 29.5 (8.7) | 13.4 (4.4) | 37.1 (8.1)

5. Secondary Outcome: Area Under the Concentration-time Curve for the Dosing Interval (AUC0-tau) for Romosozumab
Description: Area under the serum romosozumab concentration-time curve from time 0 to tau (tau = 14 days for Q2W dose cohorts and 28 days for Q4W dose cohorts)
Time Frame: as for outcome 3
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be adequately estimated.
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 5 | 6
μg*day/mL
  First dose | 65.5 (15.6) | 202 (48) | 152 (63) | 340 (73) | 71.3 (11.8) | 434 (81)
  Last dose | 141 (41) | 231 (58) | 321 (97) | 462 (97) | 136 (42) | 555 (181)

6. Secondary Outcome: Half-life Associated With the Terminal Phase of Elimination (T1/2) for Romosozumab
Time Frame: Q2W dose groups: days 71 (predose) to 169; Q24 dose groups: days 57 (predose) to 169.
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be adequately estimated.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 5 | 6
days | 7.02 (3.52) | 6.51 (1.37) | 9.32 (1.88) | 6.84 (1.79) | 6.77 (1.92) | 6.07 (1.50)

7. Secondary Outcome: Accumulation Ratio (AR) for Romosozumab
Description: The accumulation ratio (AR) was calculated as the ratio of AUC0-tau after the last dose to AUC0-tau after the first dose.
Time Frame: as for outcome 3
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be adequately estimated.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 5 | 6 | 6 | 4 | 5 | 6
ratio | 2.15 (0.45) | 1.17 (0.26) | 2.35 (0.90) | 1.35 (0.19) | 1.90 (0.49) | 1.26 (0.23)

8. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Total Spine
Description: Bone mineral density was determined by dual energy X-ray absorptiometry (DXA) scans of the lumbar spine (L1-L4) and assessed by a central lab.
Time Frame: Baseline and days 29, 85, 127, and 169
Population: Treated participants with available data at baseline and each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 29: number analyzed (Participants) | 11 | 5 | 5 | 6 | 5 | 5 | 6
  Day 29 | -0.046 (0.778) | 2.161 (0.177) | 0.541 (1.296) | -0.495 (0.930) | -0.257 (0.623) | 2.662 (0.804) | -0.660 (1.240)
  Day 85: number analyzed (Participants) | 11 | 5 | 5 | 6 | 4 | 5 | 6
  Day 85 | -0.843 (0.829) | 3.579 (1.942) | 3.881 (1.437) | 3.853 (0.543) | 3.146 (2.027) | 3.135 (1.085) | 4.157 (0.714)
  Day 127: number analyzed (Participants) | 10 | 5 | 5 | 6 | 4 | 5 | 6
  Day 127 | 0.177 (0.907) | 4.313 (3.057) | 7.219 (1.243) | 6.350 (0.732) | 5.566 (2.142) | 4.462 (1.787) | 5.599 (0.756)
  Day 169: number analyzed (Participants) | 11 | 5 | 5 | 6 | 6 | 5 | 6
  Day 169 | -0.559 (1.013) | 4.769 (1.916) | 4.835 (1.116) | 5.250 (1.630) | 4.980 (2.111) | 5.187 (0.825) | 6.560 (1.293)

9. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Total Hip
Description: Bone mineral density was determined by dual energy X-ray absorptiometry (DXA) scans and assessed by a central lab.
Time Frame: Baseline and days 29, 85, 127, and 169
Population: Treated participants with available data at baseline and each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 29: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 29 | -0.552 (0.347) | 0.528 (0.617) | -0.768 (0.334) | 0.112 (0.940) | -0.318 (1.182) | 1.244 (1.368) | -0.902 (0.408)
  Day 85: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 85 | -0.613 (0.529) | 1.066 (0.938) | 0.639 (0.608) | 2.116 (0.477) | 2.088 (0.550) | 1.134 (0.797) | 0.731 (0.621)
  Day 127: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 127 | -0.793 (0.623) | 0.702 (1.180) | 0.621 (0.940) | 2.855 (0.778) | 3.996 (1.109) | 2.111 (0.486) | 1.455 (0.669)
  Day 169: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 169 | -0.511 (0.380) | 1.423 (1.047) | 0.894 (1.013) | 3.176 (1.105) | 2.094 (0.751) | 1.007 (0.422) | 0.370 (0.629)

10. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Femoral Hip
Description: Bone mineral density was determined by dual energy X-ray absorptiometry (DXA) scans and assessed by a central lab.
Time Frame: Baseline and days 29, 85, 127, and 169
Population: Treated participants with available data at baseline and each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 29: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 29 | -0.394 (0.573) | 0.300 (0.813) | -2.172 (1.331) | -0.811 (1.596) | -0.473 (1.987) | 0.471 (1.919) | -0.597 (0.839)
  Day 85: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 85 | -1.175 (1.042) | 1.360 (1.031) | 0.578 (1.285) | -0.123 (1.001) | 0.270 (1.176) | 1.301 (0.681) | 1.956 (1.493)
  Day 127: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 127 | -2.301 (0.745) | 1.284 (1.255) | -1.005 (2.609) | 1.471 (1.228) | 1.332 (2.488) | 1.861 (1.208) | 0.091 (1.110)
  Day 169: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 169 | -0.447 (0.673) | 0.801 (1.208) | -0.672 (1.783) | 0.510 (1.103) | 2.197 (1.674) | 1.665 (1.582) | 0.116 (2.003)

11. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Distal One-third Radius
Description: Bone mineral density was determined by dual energy X-ray absorptiometry (DXA) scans and assessed by a central lab.
Time Frame: Baseline and days 29, 85, 127, and 169
Population: Treated participants with available data at baseline and each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 29: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 29 | 1.676 (0.897) | -0.220 (0.998) | -0.900 (0.733) | -2.052 (1.295) | -2.968 (0.930) | -0.435 (1.078) | -1.185 (1.101)
  Day 85: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 85 | 0.609 (0.943) | -0.082 (1.012) | -2.740 (0.770) | 0.803 (1.411) | -4.125 (0.421) | -2.504 (1.777) | -0.993 (1.478)
  Day 127: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 127 | 0.835 (0.988) | 0.680 (1.345) | -1.037 (0.668) | 0.633 (1.450) | -4.739 (0.642) | -1.756 (1.158) | -2.263 (1.227)
  Day 169: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 169 | -0.191 (0.753) | 0.522 (1.835) | 0.240 (1.068) | -0.028 (1.943) | -3.647 (0.924) | -1.836 (1.145) | -1.449 (1.106)

12. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Total Wrist
Description: Bone mineral density was determined by dual energy X-ray absorptiometry (DXA) scans and assessed by a central lab.
Time Frame: Baseline and days 29, 85, 127, and 169
Population: Treated participants with available data at baseline and each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 29: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 29 | 0.135 (0.529) | -0.552 (1.134) | -0.014 (0.591) | -0.020 (0.944) | -0.438 (1.054) | 0.757 (0.698) | 0.021 (0.479)
  Day 85: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 85 | 0.329 (0.604) | -0.063 (1.269) | -0.754 (0.533) | 0.448 (0.549) | -3.621 (1.424) | -0.306 (0.510) | 0.160 (0.296)
  Day 127: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 127 | 0.236 (0.563) | -1.134 (1.388) | 0.493 (0.792) | -0.739 (0.595) | -3.326 (1.895) | -0.914 (0.338) | -1.019 (0.647)
  Day 169: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 169 | 0.417 (0.768) | -1.102 (1.834) | -0.928 (0.717) | -0.234 (1.126) | -2.632 (1.466) | -0.378 (0.818) | -0.211 (0.619)

13. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Whole Body
Description: Bone mineral density was determined by dual energy X-ray absorptiometry (DXA) scans and assessed by a central lab.
Time Frame: Baseline and days 29, 85, 127, and 169
Population: Treated participants with available data at baseline and each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 29: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 29 | -0.391 (0.347) | 0.493 (0.580) | -1.122 (0.885) | -0.532 (0.188) | 0.521 (0.567) | -0.058 (0.387) | -0.611 (0.344)
  Day 85: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 85 | 0.103 (0.391) | 0.259 (0.642) | -0.324 (0.827) | 1.359 (0.276) | -0.151 (0.614) | 0.459 (0.271) | 0.243 (0.447)
  Day 127: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 127 | 0.000 (0.371) | -1.068 (0.357) | -0.486 (0.938) | 1.442 (0.862) | 0.513 (0.600) | 1.919 (0.839) | 0.012 (0.562)
  Day 169: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 169 | -0.352 (0.320) | 0.180 (1.143) | -0.294 (0.597) | 1.284 (0.637) | 0.801 (0.523) | 1.285 (0.264) | 0.218 (0.819)

14. Secondary Outcome: Percent Change From Baseline in Procollagen Type 1 N-terminal Propeptide (P1NP)
Time Frame: Baseline and days 2, 4, 6, 8, 15, 22, 29, 36, 43, 50 (Q2W only), 57, 58 (Q4W only), 60 (Q4W only), 62 (Q4W only), 64, 71, 72 (Q2W only), 74 (Q2W only), 76 (Q2W only), 78, 85, 99, 113, 127, 141, 155 and 169
Population: Treated participants with available data at baseline and each time point; data were not collected on days 50, 72, 74, and 76 for Q4W cohorts or on days 58, 60, or 62 for Q2W cohorts.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 2: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 2 | -4.55 (3.83) | 5.90 (4.97) | 4.37 (3.98) | 1.18 (4.35) | -0.71 (3.94) | 8.46 (6.50) | -0.64 (13.43)
  Day 4: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 4 | 0.81 (3.92) | 14.72 (5.61) | 16.32 (6.77) | 7.99 (10.60) | 9.53 (9.47) | 15.32 (7.40) | 10.72 (15.27)
  Day 6: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 6 | -5.99 (4.33) | 46.69 (7.59) | 32.85 (7.41) | 23.19 (10.40) | 32.18 (4.75) | 27.78 (7.72) | 33.83 (19.09)
  Day 8: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 8 | -1.65 (5.47) | 45.25 (8.02) | 37.14 (11.60) | 42.17 (3.90) | 69.31 (5.50) | 47.44 (12.82) | 70.63 (24.65)
  Day 15: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 15 | -0.87 (6.06) | 58.03 (11.52) | 66.12 (14.63) | 76.66 (21.28) | 103.66 (7.37) | 58.81 (12.45) | 123.92 (39.13)
  Day 22: number analyzed (Participants) | 12 | 6 | 5 | 6 | 6 | 5 | 6
  Day 22 | 0.20 (5.41) | 82.97 (21.49) | 53.76 (19.99) | 107.88 (19.52) | 117.63 (9.76) | 96.08 (13.47) | 142.64 (34.70)
  Day 29: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 29 | -0.36 (5.54) | 81.45 (20.35) | 26.35 (10.41) | 118.17 (17.03) | 74.50 (16.33) | 88.21 (11.96) | 115.09 (26.83)
  Day 36: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 36 | 5.42 (5.56) | 78.03 (21.98) | 59.50 (21.56) | 140.47 (17.70) | 103.87 (22.54) | 105.96 (14.87) | 147.40 (32.52)
  Day 43: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 43 | 2.97 (5.73) | 69.94 (20.47) | 62.16 (23.95) | 93.15 (20.34) | 129.43 (21.06) | 98.49 (17.18) | 139.62 (31.52)
  Day 50: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 50 | -12.20 (5.65) | 73.72 (23.57) |  | 128.64 (16.55) |  | 86.45 (14.88) |
  Day 57: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 57 | 1.74 (5.20) | 51.66 (20.71) | 3.28 (10.72) | 95.15 (21.45) | 77.00 (20.31) | 76.98 (12.12) | 74.16 (19.64)
  Day 58: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 6
  Day 58 | 12.47 (6.76) |  | -7.77 (9.58) |  | 54.04 (16.51) |  | 82.95 (20.45)
  Day 60: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 6
  Day 60 | 3.74 (5.80) |  | 0.47 (5.66) |  | 61.32 (17.08) |  | 85.82 (19.44)
  Day 62: number analyzed (Participants) | 6 | 0 | 5 | 0 | 5 | 0 | 5
  Day 62 | 5.62 (2.62) |  | 11.85 (9.79) |  | 64.38 (8.62) |  | 94.88 (12.29)
  Day 64: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 64 | 12.70 (12.29) | 49.88 (14.11) | 10.92 (11.34) | 65.34 (19.45) | 89.15 (12.34) | 68.67 (11.96) | 113.79 (18.18)
  Day 71: number analyzed (Participants) | 12 | 6 | 5 | 6 | 5 | 5 | 6
  Day 71 | 0.11 (2.87) | 51.25 (15.27) | 20.01 (13.17) | 88.47 (15.08) | 64.99 (21.83) | 60.58 (14.65) | 113.62 (19.09)
  Day 72: number analyzed (Participants) | 6 | 6 | 0 | 5 | 0 | 5 | 0
  Day 72 | -2.97 (4.13) | 32.99 (14.43) |  | 71.55 (7.88) |  | 63.76 (15.42) |
  Day 74: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 74 | -11.52 (6.52) | 49.16 (15.59) |  | 89.11 (15.49) |  | 71.99 (11.10) |
  Day 76: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 76 | -5.50 (6.48) | 45.95 (18.18) |  | 100.22 (18.29) |  | 78.57 (13.74) |
  Day 78: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 78 | 2.61 (5.24) | 51.59 (18.64) | 1.29 (11.31) | 77.58 (19.98) | 49.94 (17.55) | 75.17 (23.08) | 65.32 (13.57)
  Day 85: number analyzed (Participants) | 12 | 6 | 5 | 6 | 4 | 5 | 6
  Day 85 | -2.40 (3.78) | 35.64 (11.54) | -3.90 (10.10) | 79.77 (20.53) | 24.94 (9.30) | 54.06 (11.05) | 44.44 (22.42)
  Day 99: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 99 | -1.01 (4.04) | 3.21 (8.94) | -16.47 (8.68) | 31.38 (18.42) | -5.07 (13.01) | 14.97 (8.53) | 12.17 (16.53)
  Day 113: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 113 | 3.39 (5.36) | 5.15 (8.34) | -14.06 (8.68) | -4.43 (9.13) | -9.38 (12.06) | -0.83 (9.20) | -7.13 (11.60)
  Day 127: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 127 | 5.21 (6.81) | -3.26 (6.94) | -8.76 (9.73) | -9.51 (10.10) | -0.76 (17.80) | -7.63 (7.01) | -5.88 (9.47)
  Day 141: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 141 | 4.35 (4.72) | -5.75 (5.62) | -19.84 (7.87) | 2.88 (10.84) | 22.42 (16.17) | -12.85 (12.79) | -9.24 (8.87)
  Day 155: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 155 | 5.71 (4.91) | -5.45 (6.57) | -19.92 (9.17) | -0.73 (8.70) | 5.49 (22.07) | 1.76 (10.00) | -6.88 (9.24)
  Day 169 | 7.58 (7.52) | 4.79 (7.31) | -16.91 (7.34) | 1.42 (6.81) | 11.67 (11.51) | 5.78 (9.42) | -7.07 (10.52)

15. Secondary Outcome: Percent Change From Baseline in Osteocalcin
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 2: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 2 | -0.19 (2.81) | 6.61 (2.18) | -7.02 (4.56) | 4.95 (4.34) | -4.09 (6.71) | 9.53 (3.94) | -4.69 (5.12)
  Day 4: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 4 | -3.07 (2.54) | 1.17 (6.38) | -13.51 (1.88) | -21.97 (5.50) | 6.66 (6.63) | 9.13 (17.95) | -9.27 (2.61)
  Day 6: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 6 | -4.74 (2.91) | -5.55 (6.37) | -14.09 (5.65) | -0.71 (6.79) | 11.34 (6.43) | 16.14 (13.24) | -2.00 (3.09)
  Day 8: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 8 | -3.68 (3.16) | -7.13 (3.83) | -4.14 (6.29) | 22.82 (5.24) | 41.85 (29.46) | 17.92 (8.35) | -2.77 (4.06)
  Day 15: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 15 | -0.15 (2.34) | 23.55 (10.75) | 21.18 (6.94) | 33.18 (9.05) | 70.19 (15.1) | 45.22 (13.53) | 24.73 (5.35)
  Day 22: number analyzed (Participants) | 12 | 6 | 5 | 6 | 6 | 5 | 6
  Day 22 | -4.19 (2.06) | 29.99 (8.26) | 34.90 (16.55) | 57.55 (11.24) | 84.14 (12.09) | 61.18 (19.45) | 64.18 (10.17)
  Day 29: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 29 | 0.02 (2.67) | 49.44 (16.03) | 39.52 (11.33) | 81.71 (19.20) | 90.08 (7.79) | 55.58 (10.40) | 79.45 (17.12)
  Day 36: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 36 | 3.54 (2.61) | 48.91 (10.93) | 35.29 (9.36) | 76.70 (12.51) | 87.21 (16.45) | 35.55 (12.53) | 68.03 (8.81)
  Day 43: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 43 | 1.20 (2.85) | 45.46 (12.44) | 30.75 (14.39) | 77.15 (14.86) | 90.14 (17.06) | 57.62 (13.39) | 82.02 (14.92)
  Day 50: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 50 | 0.92 (5.00) | 48.63 (13.20) |  | 89.23 (18.31) |  | 52.53 (19.49) |
  Day 57: number analyzed (Participants) | 12 | 6 | 5 | 6 | 5 | 5 | 6
  Day 57 | 4.07 (2.05) | 49.28 (10.45) | -0.80 (15.19) | 70.82 (16.48) | 74.73 (8.81) | 69.16 (19.15) | 81.16 (16.26)
  Day 58: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 6
  Day 58 | 7.56 (5.24) |  | 8.12 (11.58) |  | 75.01 (14.15) |  | 75.70 (20.03)
  Day 60: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 6
  Day 60 | 0.77 (5.59) |  | 3.28 (11.15) |  | 61.68 (9.37) |  | 57.90 (19.58)
  Day 62: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 5
  Day 62 | 14.12 (3.88) |  | 2.04 (9.84) |  | 67.70 (12.26) |  | 47.72 (17.80)
  Day 64: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 64 | 6.99 (4.49) | 27.01 (9.96) | 0.57 (10.33) | 60.91 (11.91) | 70.63 (10.99) | 50.40 (22.63) | 68.64 (16.90)
  Day 71: number analyzed (Participants) | 12 | 6 | 5 | 6 | 5 | 5 | 6
  Day 71 | 1.87 (3.02) | 39.49 (12.97) | 27.96 (11.89) | 81.01 (20.69) | 77.51 (7.93) | 51.69 (16.41) | 79.70 (19.98)
  Day 72: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 72 | 5.04 (5.29) | 32.17 (9.97) |  | 95.28 (20.14) |  | 63.00 (13.12) |
  Day 74: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 74 | -5.91 (2.36) | 31.72 (10.55) |  | 60.58 (13.97) |  | 52.83 (12.14) |
  Day 76: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 4 | 0
  Day 76 | -4.13 (7.92) | 36.41 (9.63) |  | 49.94 (3.93) |  | 60.11 (16.94) |
  Day 78: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 78 | -3.86 (3.35) | 29.10 (8.42) | 12.60 (11.10) | 74.99 (13.37) | 85.53 (15.09) | 56.10 (19.30) | 89.23 (23.86)
  Day 85: number analyzed (Participants) | 12 | 6 | 5 | 6 | 4 | 5 | 6
  Day 85 | -4.37 (3.11) | 41.36 (11.92) | 19.11 (9.44) | 63.71 (11.99) | 77.23 (16.82) | 48.66 (12.49) | 81.93 (31.34)
  Day 99: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 99 | -4.97 (3.94) | 21.81 (7.95) | -9.45 (6.47) | 49.49 (16.14) | 31.98 (6.31) | 33.70 (18.41) | 30.28 (26.45)
  Day 113: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 113 | 2.57 (4.85) | 4.81 (8.41) | -11.70 (6.94) | 31.46 (10.14) | 20.24 (15.41) | 12.25 (12.11) | 6.17 (10.83)
  Day 127: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 127 | -0.34 (4.46) | 2.79 (13.64) | -13.58 (4.48) | 24.45 (15.36) | 152.92 (144.30) | 5.06 (14.88) | -3.88 (11.30)
  Day 141: number analyzed (Participants) | 11 | 6 | 6 | 5 | 4 | 5 | 6
  Day 141 | -3.80 (3.25) | -2.99 (8.22) | -25.33 (10.05) | 21.63 (8.86) | 17.25 (9.58) | 8.58 (9.20) | -4.33 (7.28)
  Day 155: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 155 | -3.51 (4.78) | -6.23 (7.52) | -21.04 (7.35) | 7.69 (8.01) | 6.85 (14.51) | -7.10 (10.56) | -11.15 (14.79)
  Day 169 | 1.25 (5.30) | -7.12 (7.84) | -20.27 (8.66) | 16.81 (12.43) | 24.60 (12.75) | 2.19 (10.84) | -13.66 (10.56)

16. Secondary Outcome: Percent Change From Baseline in Bone-specific Alkaline Phosphatase (BSAP)
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 2: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 2 | -0.07 (2.80) | -4.51 (3.09) | -8.52 (3.73) | 10.25 (3.50) | 2.22 (4.04) | 5.82 (2.73) | -0.80 (4.20)
  Day 4: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 4 | 2.16 (3.11) | -2.74 (4.96) | -4.52 (7.52) | 13.74 (3.39) | 1.15 (6.14) | 8.29 (6.28) | 6.68 (3.66)
  Day 6: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 6 | 2.26 (3.85) | 11.82 (7.95) | 7.76 (3.93) | 14.17 (2.52) | 12.59 (4.56) | 3.64 (6.40) | 6.93 (1.29)
  Day 8: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 8 | -3.30 (5.72) | 20.02 (10.24) | 9.69 (4.75) | 21.51 (6.34) | 21.87 (9.57) | 24.20 (14.92) | 20.98 (2.05)
  Day 15: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 15 | -3.26 (3.45) | 31.67 (14.36) | 31.96 (6.28) | 33.68 (8.61) | 51.97 (5.28) | 15.58 (4.69) | 46.38 (8.63)
  Day 22: number analyzed (Participants) | 12 | 6 | 5 | 6 | 6 | 5 | 6
  Day 22 | 1.23 (3.14) | 39.83 (11.04) | 37.30 (4.15) | 58.45 (14.40) | 57.66 (9.91) | 27.74 (7.34) | 61.39 (14.64)
  Day 29: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 29 | -2.04 (2.94) | 56.09 (19.29) | 36.50 (8.85) | 65.10 (14.72) | 61.66 (13.21) | 36.74 (10.53) | 35.63 (13.78)
  Day 36: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 36 | 0.04 (3.62) | 54.87 (14.40) | 28.89 (7.65) | 72.39 (12.18) | 63.55 (10.27) | 43.48 (7.98) | 34.27 (7.92)
  Day 43: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 43 | -1.93 (5.02) | 49.26 (14.03) | 39.33 (10.46) | 68.54 (12.84) | 66.74 (10.38) | 27.55 (8.68) | 52.27 (13.48)
  Day 50: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 50 | -5.81 (4.23) | 45.38 (15.81) |  | 68.67 (11.00) |  | 34.97 (10.37) |
  Day 57: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 57 | -2.15 (5.99) | 41.39 (11.28) | 38.07 (11.16) | 65.28 (9.34) | 47.38 (6.06) | 38.47 (12.18) | 44.53 (11.57)
  Day 58: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 6
  Day 58 | -2.79 (8.79) |  | 29.12 (12.18) |  | 39.33 (5.29) |  | 44.24 (13.63)
  Day 60: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 6
  Day 60 | -7.26 (5.69) |  | 18.64 (9.41) |  | 38.07 (7.47) |  | 36.75 (11.16)
  Day 62: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 5
  Day 62 | -8.41 (5.03) |  | 24.58 (10.61) |  | 38.52 (7.59) |  | 31.71 (10.53)
  Day 64: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 64 | -8.42 (5.15) | 34.60 (12.41) | 19.54 (5.71) | 77.50 (10.29) | 38.38 (7.43) | 27.78 (13.26) | 45.24 (9.78)
  Day 71: number analyzed (Participants) | 12 | 6 | 5 | 6 | 5 | 5 | 6
  Day 71 | -8.14 (4.26) | 34.29 (11.32) | 16.29 (6.39) | 52.77 (7.72) | 44.72 (9.30) | 25.46 (15.12) | 47.47 (9.99)
  Day 72: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 72 | -7.83 (3.96) | 32.18 (12.27) |  | 50.19 (10.57) |  | 19.60 (10.46) |
  Day 74: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 74 | -11.97 (7.31) | 20.46 (15.03) |  | 57.85 (10.91) |  | 15.07 (13.92) |
  Day 76: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 4 | 0
  Day 76 | -9.30 (5.16) | 40.67 (12.44) |  | 51.82 (9.53) |  | 17.91 (12.86) |
  Day 78: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 78 | -3.54 (4.26) | 33.07 (12.20) | 19.74 (6.38) | 64.46 (11.16) | 43.30 (14.16) | 13.37 (7.30) | 47.07 (12.38)
  Day 85: number analyzed (Participants) | 12 | 6 | 5 | 6 | 4 | 5 | 6
  Day 85 | -1.70 (3.61) | 26.01 (12.18) | 7.70 (5.59) | 69.90 (21.35) | 38.27 (4.20) | 18.68 (9.63) | 42.53 (14.53)
  Day 99: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 99 | -3.35 (4.67) | 23.36 (10.68) | -1.91 (3.22) | 24.89 (14.52) | 5.10 (1.62) | 17.55 (17.51) | 13.75 (6.54)
  Day 113: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 113 | 7.31 (6.57) | 10.26 (9.51) | -3.15 (3.85) | 14.75 (5.08) | -5.26 (10.20) | -6.58 (3.92) | 14.50 (5.38)
  Day 127: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 127 | 0.52 (5.26) | -2.73 (7.12) | -2.30 (4.12) | 9.62 (6.27) | 1.13 (6.36) | -6.54 (7.54) | 5.26 (5.75)
  Day 141: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 141 | 2.55 (5.44) | -1.68 (6.67) | -5.98 (5.03) | 2.90 (7.10) | 3.75 (3.96) | -4.71 (4.43) | 9.34 (3.25)
  Day 155: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 155 | 5.25 (5.28) | -0.82 (6.82) | -4.10 (4.67) | 6.15 (4.92) | 5.12 (6.77) | -4.11 (3.38) | 6.78 (8.32)
  Day 169 | 3.90 (5.22) | -1.37 (6.27) | -5.72 (5.75) | 2.33 (4.19) | 16.26 (7.56) | -4.76 (5.36) | -0.42 (6.39)

17. Secondary Outcome: Percent Change From Baseline in Serum C-telopeptide (sCTX)
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 2: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 2 | -7.31 (4.30) | 12.29 (9.15) | -11.32 (4.22) | 8.05 (9.96) | -7.07 (7.36) | -10.15 (10.74) | -6.57 (3.50)
  Day 4: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 4 | -5.51 (5.87) | 1.10 (12.49) | -19.03 (9.12) | -26.84 (4.63) | -25.85 (7.05) | -22.01 (3.66) | -34.13 (3.28)
  Day 6: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 6 | -12.60 (5.74) | -8.29 (12.56) | -26.11 (10.32) | -28.04 (7.70) | -36.98 (5.38) | -28.83 (6.44) | -35.78 (3.37)
  Day 8: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 8 | -17.79 (5.06) | -14.65 (11.02) | -31.59 (10.22) | -28.92 (3.05) | -35.93 (3.90) | -42.09 (4.09) | -43.93 (3.44)
  Day 15: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 15 | -18.86 (5.92) | -14.39 (9.41) | -35.11 (8.69) | -35.27 (4.30) | -33.00 (7.65) | -39.34 (2.85) | -48.74 (5.56)
  Day 22: number analyzed (Participants) | 12 | 6 | 5 | 6 | 6 | 5 | 6
  Day 22 | -12.98 (6.18) | -4.88 (9.99) | -29.97 (12.42) | -37.34 (3.50) | -22.85 (7.88) | -36.63 (6.67) | -39.21 (4.70)
  Day 29: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 6
  Day 29 | -10.94 (6.87) | 0.31 (6.08) | -21.11 (8.86) | -25.43 (6.08) | -21.54 (10.95) | -32.76 (4.85) | -34.53 (8.14)
  Day 36: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 36 | -20.96 (7.87) | 4.50 (11.96) | -21.42 (12.02) | -38.33 (2.21) | -29.20 (15.71) | -36.51 (9.31) | -50.32 (4.78)
  Day 43: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 43 | -14.14 (7.40) | 3.91 (9.40) | -13.79 (15.06) | -34.04 (3.35) | -20.49 (12.73) | -28.54 (6.07) | -44.64 (7.31)
  Day 50: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 50 | -12.62 (7.98) | -4.78 (11.11) |  | -26.11 (5.90) |  | -22.42 (15.96) |
  Day 57: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 57 | -17.59 (6.11) | 14.35 (10.32) | -4.53 (17.99) | -23.74 (6.45) | -13.47 (15.73) | -25.25 (12.27) | -31.52 (7.89)
  Day 58: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 6
  Day 58 | -20.27 (7.58) |  | -9.15 (9.82) |  | -9.63 (15.05) |  | -28.19 (8.64)
  Day 60: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 6
  Day 60 | -14.95 (10.06) |  | -8.80 (13.64) |  | -22.34 (16.06) |  | -28.04 (11.68)
  Day 62: number analyzed (Participants) | 6 | 0 | 5 | 0 | 5 | 0 | 5
  Day 62 | -14.01 (10.87) |  | -25.09 (10.87) |  | -21.83 (18.62) |  | -41.37 (8.69)
  Day 64: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 64 | -10.22 (7.59) | 6.59 (16.03) | -20.16 (8.81) | -20.09 (4.55) | -18.72 (14.04) | -20.03 (12.81) | -34.86 (10.25)
  Day 71: number analyzed (Participants) | 12 | 6 | 5 | 6 | 5 | 5 | 6
  Day 71 | -15.23 (5.58) | 26.63 (14.92) | -14.42 (11.82) | -18.24 (7.26) | -14.03 (13.60) | -11.02 (18.12) | -38.38 (4.37)
  Day 72: number analyzed (Participants) | 6 | 6 | 0 | 5 | 0 | 5 | 0
  Day 72 | -19.21 (6.72) | 11.70 (13.66) |  | -17.32 (7.84) |  | -8.98 (16.64) |
  Day 74: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 74 | -6.15 (8.32) | 7.40 (11.86) |  | -16.32 (6.94) |  | -9.80 (14.64) |
  Day 76: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 76 | -19.35 (5.70) | 11.70 (9.88) |  | -17.14 (9.24) |  | -17.12 (13.70) |
  Day 78: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 78 | -18.50 (6.03) | 9.18 (11.45) | -14.82 (10.85) | -17.99 (10.44) | 11.88 (21.63) | -5.24 (18.22) | -21.66 (11.50)
  Day 85: number analyzed (Participants) | 12 | 6 | 5 | 6 | 4 | 5 | 6
  Day 85 | -12.69 (5.84) | 14.95 (13.45) | 8.97 (10.90) | -13.06 (9.08) | 13.77 (22.18) | -16.89 (16.84) | -17.17 (10.09)
  Day 99: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 99 | -20.31 (5.21) | 7.45 (8.41) | -15.79 (9.03) | -7.79 (8.64) | -5.14 (17.67) | -13.22 (17.06) | -8.18 (10.80)
  Day 113: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 113 | -15.61 (6.74) | 4.66 (11.35) | -18.77 (12.28) | 0.18 (13.58) | -7.88 (13.06) | -10.06 (10.22) | -8.20 (12.19)
  Day 127: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 127 | -19.03 (5.79) | -5.63 (13.21) | -12.96 (12.78) | 0.46 (10.01) | -4.92 (18.73) | 1.68 (14.91) | -16.92 (13.00)
  Day 141: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 141 | -21.10 (6.53) | 4.86 (10.74) | -12.11 (14.71) | 1.99 (9.89) | 13.34 (14.80) | -22.48 (5.32) | -21.35 (9.69)
  Day 155: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 155 | -21.03 (5.72) | -0.02 (8.21) | -3.37 (12.01) | 7.94 (6.33) | 1.27 (14.71) | -14.43 (12.92) | -15.00 (14.96)
  Day 169 | -16.59 (6.74) | -1.13 (8.37) | -9.38 (12.56) | -0.92 (15.29) | -0.27 (10.41) | -15.61 (11.74) | -10.10 (9.54)

18. Secondary Outcome: Percent Change From Baseline in Intact Parathyroid Hormone (iPTH)
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 2: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 2 | -5.72 (4.12) | -13.34 (6.82) | -2.09 (12.69) | 7.94 (4.48) | -1.06 (5.09) | 8.68 (5.69) | -5.04 (8.62)
  Day 4: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 4 | -18.14 (2.42) | 0.35 (13.61) | 18.59 (17.92) | 2.94 (19.63) | 1.34 (10.38) | -5.59 (31.57) | -3.14 (14.09)
  Day 6: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 6 | -22.64 (5.59) | -2.67 (8.79) | 23.15 (15.52) | 8.42 (17.70) | 43.89 (18.45) | 20.35 (21.69) | -4.22 (11.74)
  Day 8: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 8 | -22.84 (5.19) | -0.20 (6.59) | 16.68 (13.79) | -7.82 (8.93) | 12.58 (13.18) | -2.24 (9.43) | 9.33 (24.92)
  Day 15: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 15 | -8.84 (5.93) | 7.31 (12.26) | 18.72 (12.98) | -10.00 (7.92) | 67.27 (35.74) | -1.40 (14.42) | 12.46 (27.05)
  Day 22: number analyzed (Participants) | 12 | 6 | 5 | 6 | 6 | 5 | 6
  Day 22 | -9.12 (4.45) | 63.58 (41.80) | 28.93 (15.69) | 0.65 (17.49) | 69.17 (22.48) | 24.27 (21.16) | 48.13 (37.16)
  Day 29: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 29 | -7.45 (6.70) | 26.13 (14.71) | 41.90 (10.87) | 34.10 (25.51) | 41.45 (17.60) | 23.91 (21.12) | 3.68 (19.02)
  Day 36: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 36 | -14.24 (4.63) | 25.21 (11.90) | 57.32 (15.99) | 22.33 (25.29) | 54.47 (18.24) | 37.99 (26.79) | 10.94 (14.70)
  Day 43: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 43 | -14.84 (5.36) | 28.17 (11.49) | 47.38 (19.72) | 23.77 (26.38) | 73.55 (22.75) | 39.90 (17.90) | 37.55 (31.09)
  Day 50: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 50 | -7.02 (9.81) | 30.25 (19.47) |  | 34.06 (31.75) |  | 41.77 (27.38) |
  Day 57: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 57 | -13.17 (6.57) | 66.13 (35.48) | 31.59 (25.03) | 26.12 (20.92) | 26.23 (13.73) | 26.14 (26.62) | 23.55 (28.82)
  Day 58: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 6
  Day 58 | -10.21 (7.73) |  | 34.80 (16.82) |  | 57.65 (25.32) |  | 24.71 (15.33)
  Day 60: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 6
  Day 60 | -8.41 (9.17) |  | 52.00 (20.18) |  | 72.18 (16.59) |  | 56.06 (31.40)
  Day 62: number analyzed (Participants) | 6 | 0 | 6 | 0 | 5 | 0 | 5
  Day 62 | -2.33 (10.30) |  | 48.83 (20.01) |  | 47.94 (18.36) |  | 37.93 (22.34)
  Day 64: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 64 | -6.40 (8.29) | 19.81 (11.29) | 62.54 (17.33) | 30.11 (13.35) | 62.07 (18.54) | 49.59 (26.25) | 64.46 (31.92)
  Day 71: number analyzed (Participants) | 12 | 6 | 5 | 6 | 5 | 5 | 6
  Day 71 | -10.38 (3.86) | 21.65 (17.69) | 40.97 (15.06) | 7.80 (17.50) | 68.44 (26.27) | 11.07 (24.13) | 15.84 (12.81)
  Day 72: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 72 | -19.26 (8.34) | 32.07 (19.22) |  | 41.99 (35.57) |  | 30.65 (17.43) |
  Day 74: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 5 | 0
  Day 74 | -9.74 (6.73) | 32.25 (25.26) |  | 21.37 (17.25) |  | 71.86 (39.62) |
  Day 76: number analyzed (Participants) | 6 | 6 | 0 | 6 | 0 | 4 | 0
  Day 76 | -8.27 (6.56) | 32.24 (14.18) |  | 2.58 (14.33) |  | 20.58 (20.98) |
  Day 78: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 78 | -16.60 (5.70) | 21.00 (14.55) | 44.03 (11.32) | 31.00 (22.68) | 56.98 (25.29) | 28.62 (13.12) | 22.73 (27.28)
  Day 85: number analyzed (Participants) | 12 | 6 | 5 | 6 | 4 | 5 | 6
  Day 85 | -3.49 (5.98) | 16.48 (11.90) | 47.95 (9.94) | -3.99 (13.52) | 24.90 (19.86) | 33.55 (22.61) | 29.25 (25.49)
  Day 99: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 99 | -20.78 (5.77) | 20.49 (13.44) | 14.08 (7.81) | 5.91 (26.94) | 12.34 (11.46) | 3.12 (12.69) | 2.69 (19.10)
  Day 113: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 113 | -7.05 (7.87) | 0.16 (12.53) | 13.91 (11.95) | -5.87 (11.21) | -10.83 (19.52) | 13.19 (18.27) | 16.73 (18.23)
  Day 127: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 127 | -12.50 (5.08) | -16.74 (7.08) | 3.14 (14.76) | -11.32 (7.81) | -7.07 (6.79) | -2.02 (17.24) | 6.96 (13.62)
  Day 141: number analyzed (Participants) | 11 | 6 | 6 | 5 | 4 | 5 | 6
  Day 141 | -16.41 (3.26) | -5.85 (9.79) | -8.33 (8.30) | -19.91 (6.71) | -4.19 (6.92) | -16.85 (13.53) | 10.80 (18.12)
  Day 155: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 155 | -15.06 (4.78) | 1.27 (8.24) | 10.09 (11.69) | -15.78 (7.72) | 17.62 (9.94) | -3.50 (10.45) | 8.76 (16.71)
  Day 169 | -9.95 (7.25) | -18.84 (7.75) | -10.08 (13.08) | -19.71 (9.00) | 30.72 (20.07) | -3.01 (10.49) | 15.09 (21.69)

19. Secondary Outcome: Percent Change From Baseline in Sclerostin
Time Frame: Baseline and days 15, 29, 43, 57, 71, 85, 99, 113, 127, 141, 155 and 169
Population: Treated participants with available data at baseline and each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percent change
  Day 15: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 5 | 6
  Day 15 | -5.6 (4.7) | 3135.6 (665.6) | 5630.4 (478.9) | 6087.5 (651.1) | 7532.4 (627.8) | 2809.3 (241.8) | 6816.0 (775.1)
  Day 29: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 29 | -3.6 (5.4) | 4068.2 (923.8) | 2335.8 (283.2) | 7713.1 (997.9) | 4993.3 (890.2) | 3904.4 (399.2) | 4573.0 (614.4)
  Day 43: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 43 | 4.4 (8.5) | 4669.2 (1119.6) | 6229.6 (475.2) | 9023.8 (1003.7) | 8471.0 (506.6) | 4613.9 (486.2) | 6486.0 (621.2)
  Day 57: number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 5 | 6
  Day 57 | 0.4 (7.2) | 5143.9 (1145.2) | 3024.9 (290.7) | 8450.2 (545.0) | 6137.5 (1319.7) | 4450.8 (471.5) | 4739.5 (660.2)
  Day 71: number analyzed (Participants) | 12 | 6 | 5 | 6 | 5 | 5 | 6
  Day 71 | -1.9 (5.7) | 4949.6 (1133.1) | 6905.1 (875.7) | 10130.3 (1041.3) | 9114.5 (812.4) | 5405.1 (667.6) | 7735.8 (949.8)
  Day 85: number analyzed (Participants) | 12 | 6 | 5 | 6 | 4 | 5 | 6
  Day 85 | -2.2 (5.8) | 4886.5 (1085.4) | 3004.2 (538.5) | 10566.4 (1667.4) | 5403.5 (1285.7) | 5254.5 (588.9) | 4873.7 (520.7)
  Day 99: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 99 | -3.5 (6.9) | 2496.0 (806.8) | 952.8 (362.7) | 6748.3 (1165.3) | 2124.2 (736.4) | 1960.4 (461.1) | 2183.7 (520.7)
  Day 113: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 113 | -7.3 (6.5) | 883.2 (397.5) | 399.4 (175.9) | 3556.2 (627.9) | 473.3 (129.2) | 395.4 (57.0) | 804.9 (257.7)
  Day 127: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 127 | 0.2 (5.8) | 364.9 (185.9) | 161.5 (67.9) | 1410.2 (273.0) | 202.6 (58.2) | 242.5 (150.0) | 311.3 (117.9)
  Day 141: number analyzed (Participants) | 11 | 6 | 6 | 6 | 4 | 5 | 6
  Day 141 | 2.1 (7.5) | 203.9 (110.6) | 84.6 (47.3) | 524.3 (109.9) | 178.2 (101.5) | 74.2 (25.5) | 128.2 (61.5)
  Day 155: number analyzed (Participants) | 12 | 6 | 6 | 6 | 4 | 5 | 6
  Day 155 | 2.6 (9.0) | 118.8 (78.9) | 57.4 (35.5) | 298.6 (67.4) | 41.0 (21.8) | 88.6 (43.3) | 48.3 (36.6)
  Day 169 | 1.9 (9.1) | 76.1 (37.7) | 40.3 (27.8) | 177.3 (37.8) | 845.3 (528.9) | 713.7 (688.9) | 16.8 (20.9)

20. Secondary Outcome: Change From Baseline in Ionized Calcium
Time Frame: Baseline and day 169 (or earlier for participants who discontinued before day 169)
Population: Treated participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
mg/dL | 0.05 (0.17) | 0.12 (0.10) | 0.06 (0.21) | -0.07 (0.18) | -0.05 (0.04) | -0.14 (0.18) | -0.06 (0.14)

ADVERSE EVENTS:
Time Frame: 169 days
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Romosozumab 1 mg/kg Q2W in Women | Romosozumab 2 mg/kg Q4W in Women | Romosozumab 2 mg/kg Q2W in Women | Romosozumab 3 mg/kg Q4W in Women | Romosozumab 1 mg/kg Q2W in Men | Romosozumab 3 mg/kg Q4W in Men
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 10/12 | 6/6 | 6/6 | 6/6 | 5/6 | 5/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Romosozumab 1 mg/kg Q2W in Women (N=6) | Romosozumab 2 mg/kg Q4W in Women (N=6) | Romosozumab 2 mg/kg Q2W in Women (N=6) | Romosozumab 3 mg/kg Q4W in Women (N=6) | Romosozumab 1 mg/kg Q2W in Men (N=6) | Romosozumab 3 mg/kg Q4W in Men (N=6)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Romosozumab 1 mg/kg Q2W in Women (N=6) | Romosozumab 2 mg/kg Q4W in Women (N=6) | Romosozumab 2 mg/kg Q2W in Women (N=6) | Romosozumab 3 mg/kg Q4W in Women (N=6) | Romosozumab 1 mg/kg Q2W in Men (N=6) | Romosozumab 3 mg/kg Q4W in Men (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OCULAR HYPERAEMIA (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
VISION BLURRED (Eye disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
COLONIC POLYP (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
GINGIVAL ULCERATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
LIP ULCERATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1
SWOLLEN TONGUE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
ASTHENIA (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
AXILLARY PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
FEELING COLD (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
INJECTION SITE BRUISING (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
INJECTION SITE DISCOMFORT (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
INJECTION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
INJECTION SITE INDURATION (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
INJECTION SITE IRRITATION (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
INJECTION SITE PAIN (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
INJECTION SITE REACTION (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
SENSATION OF FOREIGN BODY (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
VENIPUNCTURE SITE SWELLING (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
INFECTED INSECT BITE (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 3 | 2 | 1 | 0 | 2 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
VULVITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
BACK INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CARDIAC MURMUR (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HEART RATE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
ANOREXIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 1 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 1 | 0 | 1
SENSATION OF HEAVINESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 4 | 1 | 1 | 1 | 2 | 3 | 2
LETHARGY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
MULTIPLE SCLEROSIS (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
DYSURIA (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
VULVOVAGINAL BURNING SENSATION (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HAEMATOMA (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.